CLINICAL TRIAL: NCT01480830
Title: The Use of Magnetic Endoscopic Imaging for Improving Quality Indicators in Outpatient Colonoscopy
Acronym: SCOPE GUIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCT01480830
Record Dates: First submitted 2011-11-24; First posted 2011-11-29 (Estimated); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Colonoscopy
Keywords: Quality; indicators
MeSH Terms: interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard colonoscopy (No Intervention)
- Magnetic endoscopic imaging colonoscopy (Experimental)
  Interventions: Device: Magnetic Endoscopic Imaging (MEI) colonoscopy

INTERVENTIONS:
Device: Magnetic Endoscopic Imaging (MEI) colonoscopy — Colonoscopy using the Scope Guide system (Olympus Canada Inc.) by
  Arms: Magnetic endoscopic imaging colonoscopy

SUMMARY:
Colonoscopy is an important procedure for diagnosing and treating diseases of the colon. In Canada, up to 13% all colonoscopies do not examine the full colon and are therefore incomplete. Incomplete colonoscopies happen for a number of reasons but are often due to twists and turns in the colon that make the colonoscopy difficult to perform and uncomfortable for the patient.

This randomized study is being done to test a new colonoscopy system called the Scope Guide that shows an exact 3-dimensional picture of how the colonoscopy is positioned in the patient's abdomen.

We hypothesize that the use of the Scope Guide for colonoscopy will improve measures of colonoscopy quality including rate of complete examination, patient comfort, polyp detection rate, insertion time, amount of sedation required, and need for abdominal compression.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be over the age of 18 presenting for out-patient colonoscopy to the endoscopy unit at the VG Site.

Exclusion Criteria:

* Inability or unwillingness to provide written informed consent.
* Previous incomplete or difficult colonoscopy (i.e. independent indication for use of Scope Guide).
* Colonoscopist not participating in trial.
* Current pregnancy.
* Cardiac pacemaker or any other type of implantable stimulator.
* Previous colectomy, hemicolectomy, segmental colon resection, or ileocecal resection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 633 (Actual)
Dates: Start 2012-01; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Cecal intubation rate | baseline

SECONDARY OUTCOMES:
Patient comfort | baseline
Amount of sedation required | baseline
Polyp detection rate | baseline
Use of abdominal compression | baseline
Insertion time | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Donald MacIntosh, MD, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Capital District Health Authority, Halifax, Nova Scotia, Canada